CLINICAL TRIAL: NCT00534781
Title: Radiofrequency-based Plasma Microdebridement Compared to Surgical Microdebridement for Treating Achilles Tendinosis: A Prospective, Randomized, Controlled Multi-Center Study"
Brief Title: Achilles Tendinosis Study; Comparison of Radiofrequency to Surgical MicroDebridement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ArthroCare Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SM-107WW
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Achilles Pain; Achilles Tendinosis; Heel Pain
Keywords: Achilles; Tendinosis; Tendinitis; Achilles Tendinosis; Achilles Tendinitis; Coblation; Bipolar Radiofrequency; Surgical Debridement; Debridement; Heel Pain; Achilles Pain
MeSH Terms: conditions — Tendinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): plasma microtenotomy
  Interventions: Device: plasma microdebrider
- B (Active Comparator): Standard Surgical Debridement
  Interventions: Procedure: Mechanical Surgical Debridement

INTERVENTIONS:
Device: plasma microdebrider — Coblation of the Achilles
  Other Names: TOPAZ MicroDebrider
  Arms: A
Procedure: Mechanical Surgical Debridement — Surgical Debridement of the Achilles
  Arms: B

SUMMARY:
This is a research study to evaluate the outcomes after the study procedure for pain and discomfort in the heel caused from an injury in the Achilles tendon which is located on the back of the foot (commonly called "Achilles tendinitis"-Achilles tendinosis) that has not gotten better with medicine and/or other therapy.

Researchers want to see if using the study device changes outcomes for 1 year after the study procedure.

DETAILED DESCRIPTION:
Typically, Achilles pain results from overuse of the calf muscles (e.g., running, jumping) or abnormal biomechanical stress on the foot and ankle.(1). Overuse can injure the fibrous tissue that connects the heel to the calf muscles. Treating an injured Achilles tendon is crucial to avoid exacerbating the injury further, which may lead to partial or full rupture of the tendon.

Tendinosis, sometimes complicated by partial rupture, appears to be the major lesion in chronic Achilles tendinopathy; the paratenon is rarely involved. Important features are a lack of inflammatory cells and a poor intrinsic ability to heal.

Several million Americans receive treatment for tendinosis each year, with more than 200,000 patients treated each year for Achilles tendonitis and tendinosis alone.(5) Conservative treatment options for Achilles pain include rest, stretching, strengthening, ice and/or physical therapy. In general, non-surgical treatment of Achilles tendonitis and tendinosis is believed to be unsuccessful, so that surgical treatment is required in about 25% of patients; however, results of traditional surgical treatments have been reported to deteriorate with time. (3).

The purpose of this study is to evaluate longitudinal improvement of AOFAS Ankle-Hindfoot Scale scores in patients with symptomatic Achilles tendinosis treated using radiofrequency-based plasma microtenotomy compared to standard surgical debridement.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years of age
* Subject presents with pain associated with the Achilles tendon graded as >5 on a 0 to 10- point scale
* Subject's history and physical examination pinpoints anatomic origin of Achilles pain as associated with degeneration of the Achilles (non-insertional - proximal to retrocalcaneal bursa)
* Magnetic resonance imaging findings consistent with tendinosis
* Subject (or guardian) must sign IRB approved informed consent form
* Subject is willing and able to complete required follow-up

Exclusion Criteria:

* Use of NSAID's (e.g., ibuprofen, naproxen) within 2 weeks prior to treatment by this study
* Previous Achilles surgery on pathology to be treated by this study
* Heel pain associated with plantar fasciosis
* Multiple anatomic origins of pain in foot to be treated by study
* History or documentation showing Type I and Type II Diabetes Mellitus
* Physical findings and documentation of coagulopathy, infection, tumor or other systemic disease(s)
* History or documentation showing peripheral vascular disease or autoimmune disease
* Subject is currently participating in another drug/device study related to the degenerated Achilles
* Pregnant or pregnant suspected subjects prior to treatment
* History of Extracorporeal Shock Wave Treatment (ESWT) on foot to be treated by study
* Subject is incapable of understanding or responding to the study questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-09; Primary Completion 2008-07 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
To determine whether patients treated using plasma microtenotomy demonstrate equivalent longitudinal improvement of AOFAS Ankle-Hindfoot Scale scores through 12 months postoperatively to patients treated using standard surgical debridement. | 12 months

SECONDARY OUTCOMES:
To determine whether recovery from postoperative pain, quality of life and clinical events are equivalent for treatment groups. | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Terry Philbin, D.O., Principal Investigator — Orthopedic Foot and Ankle Center, Columbus, OH
Locations (2):
- United States (2):
  - Greater Chesapeake Orthopaedic Associates, Baltimore, Maryland
  - Orthopaedic Foot and Ankle Center, Columbus, Ohio

REFERENCES:
- See also: Related Info — http://topazinfo.com